CLINICAL TRIAL: NCT03180177
Title: A Phase III Multicenter Prospective Randomized Controlled Clinical Trial of HIPEC as NACT and Postoperative Chemotherapy After Interval Debulking Surgery in the Treatment of Advanced-Stage Epithelial Ovarian Cancer
Brief Title: Efficacy of HIPEC as NACT and Postoperative Chemotherapy in the Treatment of Advanced-Stage Epithelial Ovarian Cancer
Acronym: EHNPCTASEOC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shu-Zhong Cui (Other)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Henan Provincial People's Hospital (Other); Xiangya Hospital of Central South University (Other); The Third Xiangya Hospital of Central South University (Other); Peking University Cancer Hospital & Institute (Other); Peking University People's Hospital (Other); Cancer Hospital of Guizhou Province (Other); Chinese PLA General Hospital (Other); Hebei Medical University Fourth Hospital (Other); The Second Hospital of Hebei Medical University (Other); West China Second University Hospital (Other); Peking Union Medical College Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Henan Cancer Hospital (Other Government); Tianjin Medical University Cancer Institute and Hospital (Other); The Third Affiliated Hospital of Guangzhou Medical University (Other); Wuhan University (Other); RenJi Hospital (Other); Obstetrics & Gynecology Hospital of Fudan University (Other); Southern Medical University, China (Other); Fourth Affiliated Hospital of Guangxi Medical University (Other); Shandong Cancer Hospital and Institute (Other); Beijing Obstetrics and Gynecology Hospital (Other); Chongqing Cancer Institute (Unknown); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Xinqiao Hospital of Chongqing (Other)
Responsible Party: Sponsor-Investigator, Shu-Zhong Cui, President of Affiliated Tumor Hospital of Guangzhou Medical University, Affiliated Cancer Hospital & Institute of Guangzhou Medical University
Organization: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIPEC-03
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Epithelial Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
Keywords: Hyperthermic Intraperitoneal Chemotherapy; Neoadjuvant Chemotherapy; Interval Debulking Surgery; Advanced-Stage Epithelial Ovarian Cancer; Postoperative Chemotherapy
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy; Neoadjuvant Therapy; Chemotherapy, Adjuvant

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 1. Hyperthermic Intraperitoneal Chemotherapy (HIPEC) with paclitaxel 175 mg/m^2 and cisplatin 75 mg/m^2 intraperitoneally in succession
  2. 2 cycles of neoadjuvant chemotherapy: paclitaxel 175 mg/m^2 IV>3 hour+ carboplatin AUC = 5-6 IV>1 hour, every 3 weeks
  3. Interval debulking surgery
  4. Hyperthermic Intraperitoneal Chemotherapy (HIPEC) with paclitaxel 175 mg/m^2 and cisplatin 75 mg/m^2 intraperitoneally in succession
  5. 2 cycles of adjuvant chemotherapy: paclitaxel 175 mg/m^2 IV>3 hour+ carboplatin AUC = 5-6 IV>1 hour, every 3 weeks
  Interventions: Procedure: Hyperthermic Intraperitoneal Chemotherapy; Procedure: Interval debulking surgery; Drug: neoadjuvant chemotherapy; Drug: adjuvant chemotherapy
- Control group (Active Comparator): 1. 3 cycles of neoadjuvant chemotherapy: paclitaxel 175 mg/m^2 IV>3 hour+ carboplatin AUC = 5-6 IV>1 hour, every 3 weeks
  2. Interval debulking surgery
  3. 3 cycles of adjuvant chemotherapy: paclitaxel 175 mg/m^2 IV>3 hour+ carboplatin AUC = 5-6 IV>1 hour, every 3 weeks
  Interventions: Procedure: Interval debulking surgery; Drug: neoadjuvant chemotherapy; Drug: adjuvant chemotherapy

INTERVENTIONS:
Procedure: Hyperthermic Intraperitoneal Chemotherapy — HIPEC is performed as neoadjuvant chemotherapy(NACT) and postoperative chemotherapy after interval debulking surgery (IDS) for advanced-stage epithelial ovarian cancer. The first HIPEC is conducted within 24h after laparoscopic exploration or Interval debulking surgery: Paclitaxel 175 mg/m^2, 43°C, 90min. The second HIPEC is performed after 48 hours of the first HIPEC. The second HIPEC regimens are cisplatin 75 mg/m^2, 43°C, 90min.
  Other Names: HIPEC
  Arms: Experimental group
Procedure: Interval debulking surgery — Cytoreductive surgery (CRS) is performed after neoadjuvant chemotherapy.
  Other Names: IDS
Drug: neoadjuvant chemotherapy — Systemic chemotherapy regimens after HIPEC treatment are paclitaxel 175 mg/m^2 IV>3 hour+ carboplatin AUC = 5-6 IV>1 hour, every 3 weeks for 2 cycles in experimental group.
  Systemic chemotherapy regimens after laparoscopic exploration are paclitaxel 175 mg/m^2 IV>3 hour+ carboplatin AUC = 5-6 IV>1 hour, every 3 weeks for 3 cycles in control group.
  Other Names: NACT
Drug: adjuvant chemotherapy — Systemic chemotherapy regimens after HIPEC treatment are paclitaxel 175 mg/m^2 IV>3 hour+ carboplatin AUC = 5-6 IV>1 hour, every 3 weeks for 2 cycles in experimental group.
  Systemic chemotherapy regimens after IDS are paclitaxel 175 mg/m^2 IV>3 hour+ carboplatin AUC = 5-6 IV>1 hour, every 3 weeks for 3 cycles in control group.
  Other Names: ACT

SUMMARY:
This project is a multi-center, prospective, randomized controlled clinical observation the safety and efficacy of hyperthermic intraperitoneal chemotherapy as neoadjuvant chemotherapy(NACT) and postoperative chemotherapy after interval debulking surgery (IDS) for advanced-stage epithelial ovarian cancer . PR/SD rate, percentage of optimal debulking surgery and 3-year disease-free survival is the primary end points of this project.

DETAILED DESCRIPTION:
The current standard treatment for epithelial ovarian cancer, tubal cancer, and primary peritoneal cancer is maximal cytoreductive surgery followed by intravenous chemotherapy with or without intraperitoneal chemotherapy (IP). Recently, the organizations of SGO and ASCO recommended that women with a high perioperative risk profile or a low likelihood of achieving cytoreduction to < 1 cm of residual disease (ideally to novisible disease) should receive neoadjuvant chemotherapy.

Hyperthermia promotes chemotherapy to penetrate deeper into the cancer tissue. Therefore, hyperthermic intraperitoneal chemotherapy (HIPEC) as neoadjuvant chemotherapy and postoperative chemotherapy after interval debulking surgery in the treatment of ovarian cancer could lead to higher response rate and better survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Disease status primary epithelial ovarian cancer, tubal cancer, and primary peritoneal cancer (Stage III and IV)
* Fagotti score by laparoscopic exploration >= 6
* After receiving HIPEC+neoadjuvant chemotherapy (NACT) or NACT alone, the curative effects evaluated according to RICIST criteria is partial remission (PR) and stable disease (SD).
* Residual tumor < 1cm after completion of interval debulking surgery
* 18 < Age < 70 year old
* Expected survival > 3 months
* Performance status: ECOG 0-1
* Adequate bone marrow function Hb ≥8 g/dl (After correction in case of iron deficient anemia) WBC ≥ 3,000/mm3, Platelet ≥ 100,000/mm3
* Adequate renal function Creatinine ≤ 1.5 mg/dl, and adequate hepatic function Bilirubin ≤ 1.5 mg/dl and AST and ALT ≤ 80 IU/L
* Voluntary participation after getting written informed consent.

Exclusion Criteria:

* Fagotti score by laparoscopic exploration < 6
* After receiving HIPEC+neoadjuvant chemotherapy (NACT) or NACT alone, the progression of disease (PD) is evaluated by doctor.
* Suboptimal debulking (residual tumor > 1cm)
* Extensive adhesion in peritoneal cavity
* Previous History of other malignancies (except excision of skin cancer, thyroid cancer)
* Poorly controlled disease e.g. atrial fibrillation, stenocardia, cardiac insufficiency, persistent hypertension despite medicinal treatment, ejection fraction<50%
* Receiving other chemotherapy, radiotherapy or immunotherapy
* Patients who are unsuitable candidates by doctor's decision
* Without given written informed consent

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
PR/SD rate | Through study completion, an average of 1 year
  calculate the percent of partial remission (PR) plus stable disease (SD) of patients received HIPEC+NACT or NACT alone in both two arms
Percentage of optimal debulking surgery | Through study completion, an average of 1 year
  evaluate the percentage of optimal debulk (residual disease < 1cm) after interval debulking surgery between study arms
Disease-free survival rate | 3 years
  assess disease free survival rate during 3 years in both study arms

SECONDARY OUTCOMES:
Overall survival rate | 3 years
  assess overall survival rate during 3 years in both study arms
Risk factors for morbidity and mortality | Through study completion, an average of 1 year
  determine percent of patients wtih Grade I-IV adverse events according to NCI criteria, Common Terminology Criteria for AE (CTCAE 4.0).
Quality of life | 3 years
  Evaluated according to European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Cancer (EORTC QLQ-C30)
Quality of life for ovarian cancer | 3 years
  Evaluated according to European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Ovarian Cancer Module (QLQ-OV28)

CONTACTS AND LOCATIONS:
Overall Officials: Shuzhong Cui, M.D, Study Director — Affiliated Cancer Hospital & Institute of Guangzhou Medical University; Zhongqiu Lin, M.D, Study Director — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Department of Abdominal Surgery (Section 2), Affiliated Tumor Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No